CLINICAL TRIAL: NCT03468946
Title: Investigation of the Relationship Between Taste Perception and Caries Activity in School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Edibe Egil, Assistant Professor, University of Beykent
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: SAG-C-DRP-090414-0077
Record Dates: First submitted 2018-02-19; First posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Healthy
Keywords: taste perception; caries risk; cariogram; children
MeSH Terms: interventions — Sodium Chloride; Caffeine; Citric Acid; Candy; Sucrose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high caries risk (Other): children with high caries -identified by cariogram to evaluate sweet taste perception, salty taste perception, sour taste perception and bitter taste perception of school children and compare them with demographic, clinical, microbiologic and biochemical caries-risk factors.
  Interventions: Other: salty taste perception; Other: bitter taste perception; Other: sour taste perception; Other: sweet taste perception
- medium caries risk (Other): children with medium caries- identified by cariogram to evaluate sweet taste perception, salty taste perception, sour taste perception and bitter taste perception of school children and compare them with demographic, clinical, microbiologic and biochemical caries-risk factors.
  Interventions: Other: salty taste perception; Other: bitter taste perception; Other: sour taste perception; Other: sweet taste perception
- low risk (Other): no caries or low risk- identified by cariogram to evaluate sweet taste perception, salty taste perception, sour taste perception and bitter taste perception of school children and compare them with demographic, clinical, microbiologic and biochemical caries-risk factors.
  Interventions: Other: salty taste perception; Other: bitter taste perception; Other: sour taste perception; Other: sweet taste perception

INTERVENTIONS:
Other: salty taste perception — salty taste perception in high caries risk, medium caries risk, low caries risk.
  The aim of this study was to evaluate salty taste perceptions of school children and compare them with demographic, clinical, microbiologic and biochemical caries-risk factors(high caries risk, medium caries risk, low risk ).
  Other Names: sodium chloride; Sigma-Aldrich, USA; RIEDEL SK.S.314
Other: bitter taste perception — bitter taste perception in high caries risk, medium caries risk, low caries risk.
  The aim of this study was to evaluate bitter taste perceptions of school children and compare them with demographic, clinical, microbiologic and biochemical caries-risk factors (high caries risk, medium caries risk, low risk ).
  Other Names: caffeine; Merck, Germany; MERCK 102584
Other: sour taste perception — sour taste perception in high caries risk, medium caries risk, low caries risk. The aim of this study was to evaluate sour taste perceptions of school children and compare them with demographic, clinical, microbiologic and biochemical caries-risk factors (high caries risk, medium caries risk, low risk ).
  Other Names: citric acid; Sigma-Aldrich, USA; RIEDEL SK.R.2 7102
Other: sweet taste perception — sweet taste perception in high caries risk, medium caries risk, low caries risk.
  The aim of this study was to evaluate sweet taste perceptions of school children and compare them with demographic, clinical, microbiologic and biochemical caries-risk factors (high caries risk, medium caries risk, low risk ).
  Other Names: sucrose; Merck, Germany; MERCK 1.07651.1 000

SUMMARY:
Four basic taste perceptions and relationship with caries are poorly investigated in children as compared to adults.

The aim of this study was to evaluate salty, sweet, bitter and sour taste perceptions of school children and compare them with demographic, clinical, microbiologic and biochemical caries-risk factors.

DETAILED DESCRIPTION:
Study design

1. Caries risk assessment The investigators developed a questionnaire to understand the patient's overall health status, to collect demographic and socio-economic information, to assess their oral health habits. The questionnaire consists of 3 parts; first part includes questions about general health such as chronic diseases, drugs and allergies, second part includes questions about income and education level of parents, and last part includes questions about oral health knowledge, habits, diet contents and frequency, fluoride exposure. the investigators allowed the parents to fill the questionnaire.

   After the questionnaire was filled, the investigators performed the oral examination using DMFT, DMFS, dft and dfs indices according to WHO. Then, the investigators determined the oral hygiene status with Sillness&Löe Index (Silness ve Loe, 1964). the investigators estimated paraffin-stimulated salivary flow rate, buffer capacity, mutans streptococci and lactobacilli counts using CRT chairside kits (Ivoclar Vivadent, Schaan, Liechtenstein).

   In addition to initial questionnaire and oral examination, the investigators asked the patients to record their nutritional takings of 2 weekdays and 1 weekend day. the investigators estimated the caries risk profiles of all children using the Cariogram which is a computer-based program. Cariogram identifies three risk groups low, medium and high caries risk according the scores.
2. Taste evaluation the investigators prepared aqueous basic taste solutions of sucrose (Merck, Germany, purity >99.5%), sodium chloride (Sigma-Aldrich, USA, purity >99%), caffeine (Merck, Germany, purity >99.5%), citric acid monohydrate (Sigma-Aldrich, USA, purity >99%), at two levels (1.0 ISO, 2.0 ISO) (ISO 3972:1991, 8586-1:1993) (Table 1). the investigators formulated all the solutions by using spring water in the same day of measurement at room temperature (25 ± 2°C). Each solution was coded randomly.

ELIGIBILITY:
Inclusion Criteria:

- without any chronic disease such as diabetes and being ASA I or ASA II. We only included patients who had no antibiotics and drug intake within the last month.

Exclusion Criteria:

- chronic disease ASA III, IV antibiotic and drug intake within the last month

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2013-05-02 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
DMFT, DMFS, dft and dfs indices | 1 year
  DMFT, DMFS, dft and dfs indices are total counts of decayed, missing, filled teeth / DMFT, Plaque index, Salivary flow rate, buffer capacity, mutans streptococci and lactobacilli counts are combined to report caries risk in high/medium/low caries risk

SECONDARY OUTCOMES:
Sillness&Löe Index | 1 year
  Sillness&Löe index in total amount of dental plaque on the teeth. /DMFT, Plaque index, Salivary flow rate, buffer capacity, mutans streptococci and lactobacilli counts are combined to report caries risk in high/medium/low caries risk
Salivary flow rate | 1 year
  Salivary flow rate in ml/minute
buffer capacity | 1 year
  buffer capacity in pH / DMFT, Plaque index, Salivary flow rate, buffer capacity, mutans streptococci
mutans streptococci and lactobacilli counts | 1 year
  mutans streptococci and lactobacilli counts in cfu/ml / DMFT, Plaque index, Salivary flow

IPD SHARING:
Plan to Share IPD: No